CLINICAL TRIAL: NCT05967234
Title: THIS-WIC Vermont Breastfeeding Education Application Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Vermont WIC (Unknown); RTI International (Other)
Responsible Party: Principal Investigator, Erin Hennessy, Assistant Professor, Division of Nutrition Interventions, Communication and Behavior Change Director ad interim, ChildObesity180 Friedman School of Nutrition Science and Policy, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB # 308
Record Dates: First submitted 2023-06-06; First posted 2023-08-01 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Telehealth; Breast Feeding; WIC
Keywords: Telehealth; WIC; Breast feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Study participants will be clients at local WIC agency sites where the telehealth solution is offered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth solution (Experimental): Telehealth solution offered for breastfeeding education.
  Interventions: Behavioral: Telehealth solution

INTERVENTIONS:
Behavioral: Telehealth solution — Telehealth solution offered for breastfeeding education.

SUMMARY:
With funding through USDA and Tufts University's Telehealth Intervention Strategies for WIC (THIS-WIC) project, the Vermont WIC department will be conducting a feasibility study of a mobile telehealth solution for breastfeeding education. The purpose of this study is to evaluate this telehealth solution. The research/evaluation involves completing online surveys and interviews. The evaluation will focus on participant satisfaction, usage of the telehealth solution, and use of information collected on WIC participant through the WIC management information system (MIS) and the telehealth platform. It is hypothesized that the telehealth solution will increase WIC participant's satisfaction with breastfeeding education.

DETAILED DESCRIPTION:
Telehealth can reduce barriers and increase access to care, and it can be applied to the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC). WIC is a federal nutrition assistance program that helps low-income women with children up to age 5. There is a large volume of research that supports remote patient monitoring, and the most benefits are found when telehealth is used for communication and counseling. The USDA awarded Tufts University a grant to test and evaluate the use of telehealth innovations in the delivery of USDA's WIC program. Tufts University then offered the USDA/Tufts Telehealth Intervention Strategies for WIC (THIS-WIC) grant opportunity to WIC state agencies across the US. THIS-WIC selected 7 WIC State Agencies to receive grants, and the Vermont state agency is one recipient. The THIS-WIC team at Tufts University is leading the evaluation of these telehealth solutions in collaboration with funded WIC State Agencies.

THIS-WIC aims to generate evidence from Vermont's telehealth solution to inform how the telehealth platform supports WIC services . Evaluation findings will inform stakeholders about the platform's benefits and how viable it is to sustain and adapt more widely.

The purpose of this study is to evaluate the effectiveness of this telehealth solution by having clients complete surveys and interviews on their comfortability using telehealth and their satisfaction with the telehealth solution. Additionally, information about usage will be collected from the telehealth platform, and secondary demographic and other nutrition-related information about study participants is already collected in the MIS and will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and reads English (as the telehealth solution is available in English)
* Pregnant or postpartum
* Has access to a smart phone or smart device (e.g. iPad or tablet)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the telehealth solution | During the study period, approximately 12 months
  WIC clients satisfaction with breastfeeding education offered via the telehealth solution. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.

SECONDARY OUTCOMES:
Frequency of use of the telehealth solution | During the study period, approximately 12 months
  The frequency with which WIC clients use the telehealth solution. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Intent to breastfeed | During the study period, approximately 12 months
  WIC clients intent to breastfeed. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Breastfeeding duration | During the study period, approximately 12 months
  Duration of breastfeeding in clients offered the telehealth solution. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Attitudes to breastfeeding | During the study period, approximately 12 months
  Impact of the telehealth solution on WIC clients' attitudes to breastfeeding. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Barriers encountered in use of the telehealth solution and breastfeeding | During the study period, approximately 12 months
  Barriers encountered by WIC clients in use of the telehealth solution and in breastfeeding. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hennessy, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Tufts Telehealth Intervention Strategies for WIC (THIS-WIC) — https://thiswic.nutrition.tufts.edu/